CLINICAL TRIAL: NCT02139215
Title: A Phase IV Multicenter Trial to Evaluate Real-world Health Outcomes and Economic Impact of Panitumumab Versus Standard-of-care in the Treatment of Patients With Chemotherapy-refractory Metastatic Colorectal Cancer
Brief Title: Study to Evaluate Real-world Pharmacoeconomics of Panitumumab in Metastatic Colorectal Cancer Patients
Status: Completed | Type: Observational
Sponsor: PeriPharm (Other)
Collaborators: Personalized Medicine Partnership for Cancer (Other)
Responsible Party: Sponsor
Other Study IDs: PMPC-01
Record Dates: First submitted 2014-05-13; First posted 2014-05-15 (Estimated); Last update posted 2018-03-30 (Actual); Status verified 2018-03

CONDITIONS: Colorectal Cancer Metastatic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
This is a phase IV multicenter trial to evaluate real-world health outcomes and economic impact of panitumumab versus standard-of-care (SOC) in the treatment of patients with chemotherapy-refractory metastatic colorectal cancer (mCRC).

The study will enable real-life health economics and outcome research (HEOR) to assess the impact of panitumumab in the Quebec population.

The primary objective is to evaluate real-world health outcomes and economic impact of panitumumab in the treatment of patients with chemotherapy-refractory mCRC in comparison with SOC. The secondary objectives are to confirm survival data, to assess the quality of life of patients and to assess the health care resource utilization of patients.

Patients with a mutated KRAS gene will be treated with standard-of-care (SOC) and patients with a non-mutated (wild type) KRAS gene will be treated with panitumumab.

During the course of the study, data will be collected on quality of life and work productivity. Patients will be asked to fill a set of questionnaires at their recruitment in the study and at every 3 months after treatment initiation.

ELIGIBILITY:
Inclusion Criteria:

* Patients with a histologically confirmed diagnosis of mCRC.
* Immunohistochemical evidence of EGFR expression.
* ECOG performance status of 0, 1 or 2.
* Patients refractory to fluoropyrimidine, oxaliplatin, and irinotecan chemotherapy regimens
* Patients with a wt KRAS scheduled to receive panitumumab as a single agent for the third-line treatment of mCRC or patients with a mt KRAS scheduled to receive SOC for third-line treatment of mCRC.
* Signed and dated IRB-approved informed consent document.
* Ability to read and understand English or French.
* 18 years of age or older.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with chemotherapy-refractory metastatic colorectal cancer from participating hospitals in Quebec.
Sampling Method: Non-Probability Sample
Enrollment: 72 (Actual)
Dates: Start 2014-04; Primary Completion 2018-03 (Actual); Study Completion 2018-03 (Actual)

PRIMARY OUTCOMES:
The pharmacoeconomic impact of panitumumab for the treatment of metastatic colorectal cancer in a real-life setting | From the date of registration until date of death from any cause, assessed up to 38 months
  Pharmacoeconomic impact (cost-effectiveness and cost-utility) will be evaluated by questionnaires completed by the patient and caregiver. These include quality of life, health resource utilization, work productivity and activity impairment, and health questionnaires.

CONTACTS AND LOCATIONS:
Overall Officials: Jean Lachaine, PhD, Principal Investigator — PeriPharm
Locations (5):
- Canada (5):
  - CSSS Alphonse-Desjardins (CHAU, Hôtel-Dieu de Lévis), Lévis, Quebec
  - CIUSSS de l'Est-de-l'Île-de-Montréal (Hôpital Maisonneuve-Rosemont), Montreal, Quebec
  - Centre Hospitalier de l'Université de Montréal (CHUM), Montreal, Quebec
  - Centre Hospitalier Universitaire de Sherbrooke (CHUS), Sherbrooke, Quebec
  - Centre Hospitalier Universitaire de Québec (CHU, Hôtel-Dieu de Québec), Québec